CLINICAL TRIAL: NCT01586975
Title: Multiphase Study to Determine if Platelet Function Analysis Results Correlate With Ischemic Events and Bleeding Complications
Brief Title: Aspirin Resistance and Stroke Risk: Platelet Function Analysis in Patients With Ischemic Events
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Aspirin Resistance and Stroke; IRB#0996-007 FUND#7810 (Other: Northwestern Memorial Hospital)
Record Dates: First submitted 2011-08-03; First posted 2012-04-27 (Estimated); Results first posted 2015-12-03 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Stroke; Myocardial Infarctions
MeSH Terms: conditions — Stroke; Myocardial Infarction | interventions — Clopidogrel; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Clopidogrel 75 mg (Active Comparator): Clopidogrel 75 mg daily
  Interventions: Drug: Clopidogrel
- Aspirin 81 mg (Active Comparator): open-label Aspirin 81 mg daily
  Interventions: Drug: Aspirin 81 mg
- Aspirin > 300mg (Active Comparator): open-label Aspirin over 300 mg daily
  Interventions: Drug: Aspirin >300 mg

INTERVENTIONS:
Drug: Clopidogrel — Clopidogrel 75 mg QD
  Other Names: Plavix
  Arms: Clopidogrel 75 mg
Drug: Aspirin 81 mg — Aspirin 81mg QD
  Other Names: Acetylsalicylic Acid; ASA
  Arms: Aspirin 81 mg
Drug: Aspirin >300 mg — Aspirin >300 mg QD
  Other Names: Acetylsalicylic Acid; ASA
  Arms: Aspirin > 300mg

SUMMARY:
The purpose of this study is to determine if PFA results correlate with ischemic event outcomes as well as bleeding complications. Hypothesis is antiplatelet agents will be more efficacious if they are administered in a dose-adjusted manner using PFA results as a guide.

DETAILED DESCRIPTION:
Atherothrombotic disease is a leading killer of adults throughout the world. The current mainstay for the prevention of ischemic vascular events is the use of aspirin Antiplatelet agents are used routinely for the primary and secondary prevention of vascular events in patients with a prior history of stroke, TIA, or at high risk for the development of cerebrovascular disease. Numberous individual studies and meta-analyses have shown that essentially all of the oral antiplatelet agents have limited efficacy, with relative risk reductions in the range of 20-35%. The purpose of this study is to perform serial platelet function assays (PFAs) on patients with cerebrovascular disease who are taking antiplatelet agents and perform a pilot study to determine the feasibility of administering ASA as a dose adjusted medication using PFA. The long term goal of this study is to determine whether antiplatelet therapy will be more efficacious and/or safer if it is administered in a dose-adjusted manner.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be taking Aspirin or Plavix
* Patient must have had a stroke, TIA or cerebrovascular disease

Exclusion Criteria:

-None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2007-07; Primary Completion 2010-04 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Alberts, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Background] Taylor TN, Davis PH, Torner JC, Holmes J, Meyer JW, Jacobson MF. Lifetime cost of stroke in the United States. Stroke. 1996 Sep;27(9):1459-66. doi: 10.1161/01.str.27.9.1459. PMID 8784113

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with cerebrovascular disease and taking one or more antiplatelet medication were consented for study participation from 2007 though 2010. Patients were recruiting on the inpatient stroke unit at Northwestern Memorial Hospital and seen in the outpatient stroke clinic.
Groups:
- Clopidogrel 75 mg: Clopidogrel 75 mg QD
- Aspirin 81 mg: Aspirin 81 mg QD
- Aspirin > 300 mg: Aspiring > 300 mg QD
Period: Overall Study
Arm/Group | Clopidogrel 75 mg | Aspirin 81 mg | Aspirin > 300 mg
Started | 15 | 32 | 46
Completed | 15 | 32 | 46
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Aspiring >300 mg: Aspirin >300 mg QD
- Total: Total of all reporting groups
Arm/Group | Clopidogrel 75 mg | Aspirin 81 mg | Aspiring >300 mg | Total
Number analyzed (Participants) | 15 | 32 | 46 | 93
Age, Customized [Mean (Full Range); unit: years] | 60.6 [37 to 83] | 67.4 [36 to 93] | 56.2 [21 to 87] | 60.7 [21 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 16 | 26 | 51
  Male | 6 | 16 | 20 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 4 | 7 | 13
  White | 13 | 25 | 37 | 75
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 15 | 32 | 46 | 93

OUTCOME MEASURES:

1. Primary Outcome: PFA1
Description: Platelet Function Analysis (PFA) lab results: PFA was performed using the PFA 100 device (Dade-Behring), which uses a higher sheer stress flow cytometry paradigm to measure the time in seconds to closing of an aperture. Normal is defined as <172 seconds."
Time Frame: 3-6 months (Collected once between regulalary scheduled follow-up visit between 3-6 months)
Measure: Mean (Standard Error); unit: seconds
Groups:
- Aspirin 81 mg: open label Aspirin
- Aspirin > 300 mg: open-label Aspirin
Arm/Group | Clopidogrel 75 mg | Aspirin 81 mg | Aspirin > 300 mg
Number analyzed (Participants) | 15 | 32 | 46
seconds | 202.0 (27.1) | 271.1 (14.9) | 234.7 (13.4)
Statistical Analysis 1: Comparison: Clopidogrel 75 mg vs Aspirin 81 mg vs Aspirin > 300 mg; Kruskal-Wallis non-parametric ANOVA test; Test type: Superiority or Other; p = 0.0742, Kruskal-Wallis — p-value is not adjusted, and no a priori threshold was used

ADVERSE EVENTS:
Time Frame: Patients were monitored via routine clinic/office visits to determine if they had an ischemic vascular event or hemorrhagic event. These follow-up visits were scheduled every 3-6 months as per their regularly scheduled clinic follow-up visits.
Arm/Group | Clopidogrel 75 mg | Aspirin 81 mg | Aspirin >300 mg
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/32 | 2/46
Other Adverse Events (participants affected / at risk) | 2/15 | 3/32 | 2/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clopidogrel 75 mg (N=15) | Aspirin 81 mg (N=32) | Aspirin >300 mg (N=46)
Clinical Stroke (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) — one patient suffered a clinical stroke
MI (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — one patient suffered a MI
TIA (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) — one patient suffered from a TIA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clopidogrel 75 mg (N=15) | Aspirin 81 mg (N=32) | Aspirin >300 mg (N=46)
Nose bleeds (Vascular disorders) | 0 (0) | 2 (2) | 2 (2) — 4 patients suffered from nose bleeds
Bruising (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) — minor bruising
GI bleeding (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) — minor GI bleeding/blood in stool

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No